CLINICAL TRIAL: NCT01096888
Title: FFit Moms- an Internet-based Postpartum Weight Loss Program
Brief Title: Fit Moms- an Internet-based Postpartum Weight Loss Program
Acronym: FM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Women Infants and Children program WIC (Unknown)
Responsible Party: Principal Investigator, Suzanne Phelan, Principal Investigator, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CP-FM
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Postpartum Weight
Keywords: WIC; Weight loss; Overweight; Post Partum; Internet based weight loss intervention for Mothers in the WIC program.
MeSH Terms: conditions — Weight Loss; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard WIC care (No Intervention): Patients randomized to this group will receive standard WIC care and an information packet surround healthy eating and activity topics.
- Enhanced WIC weight loss program (Active Comparator): Participants randomized into this condition will receive standard WIC care, but will also receive weight loss classes provided through the internet. Topics will cover behavioral weight loss topics, based off the protocols of the Look AHEAD program.
  Interventions: Behavioral: Enhanced WIC Program

INTERVENTIONS:
Behavioral: Enhanced WIC Program — Applying an internet based weight loss intervention to participants in the WIC program to enhance weight loss post partum.
  Arms: Enhanced WIC weight loss program

SUMMARY:
The purpose of this study is to provide weight loss interventions for Mothers participating in the WIC program, using the internet to deliver weight loss materials.

DETAILED DESCRIPTION:
Develop recruitment methods and determine feasibility of recruiting WIC postpartum women who meet inclusion criteria. We will collect data on number of individuals screened and reasons for exclusions. Establish and examine feasibility and effectiveness of protocol for WIC counselors reinforcing adherence to web based program. We will assess frequency with which WIC counselors adhere to protocol of reinforcing adherence to web-based program and extent to which any "treatment contamination" occurs between WIC counselors and Standard Care participants.In those randomized to Enhanced WIC + Internet-based postpartum program, examine acceptability, burden, ease of use, frequency of technical problems, and adherence to web-based program (number of logins, message board postings)Explore whether the Enhanced WIC plus Internet postpartum weight loss program will produce significantly greater weight losses than Standard WIC at 2 months. Explore whether Enhanced WIC plus Internet postpartum weight loss program will result in greater improvements in eating and exercise behaviors (examined at 0, and 2 months) and psychosocial parameters (i.e., depression, social support, self-efficacy, body image) than standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years.
* Delivery within 6-52 weeks
* Exceed pre-pregnancy weight by at least 6.8 kg (15 pounds)
* Current BMI > 22
* English speaking
* Has computer with internet access
* Literacy of at least 5th grade reading level

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Relocating in the next year
* Serious medical problem (i.e. heart disease, cancer, renal disease and diabetes), for which physician supervision of diet and exercise prescription is needed.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Enhanced WIC program to instigate weight loss | 3 months
  We are taking the standard WIC care for Mothers who are at least 6 months post partum and enhancing their program to include an internet based weight loss intervention.

SECONDARY OUTCOMES:
Baseline characteristics that moderate the efficacy of the intervention. | 3 months
  To examine the relationship between changes in behaviors, psychosocial factors, and weight changes during the 3-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD., Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States